CLINICAL TRIAL: NCT01808638
Title: A PHASE Ib/IIa STUDY OF COMBINATION THERAPY WITH GEMCITABINE AND ATU027 IN SUBJECTS WITH LOCALLY ADVANCED OR METASTATIC PANCREATIC ADENOCARCINOMA
Brief Title: Atu027 Plus Gemcitabine in Advanced or Metastatic Pancreatic Cancer (Atu027-I-02)
Acronym: Atu027-I-02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Silence Therapeutics GmbH (Industry)
Collaborators: Granzer Regulatory Consulting & Services (Other); FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Atu027-I-02; 2012-004429-26 (EudraCT Number)
Record Dates: First submitted 2013-03-04; First posted 2013-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Adenocarcinoma; Pancreas; Gemcitabine; Atu027
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Adenocarcinoma | interventions — Atu027; Gemcitabine; Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lead in safety period (Other): Cohort of three subjects with non-pancreatic cancer for whom conventional treatment options have failed, will be treated. If one of the subjects in the safety cohort experiences an unacceptable toxicity, the safety cohort is expanded to six subjects.
  Interventions: Drug: Atu027 & gemcitabine in lead in safety period
- Treatment arm 1 (Experimental): Subjects with advanced pancreatic cancer will be treated.
  Interventions: Drug: Atu027 & gemcitabine in treatment arm 1
- Treatment arm 2 (Experimental): Subjects with advanced pancreatic cancer will be treated.
  Interventions: Drug: Atu027 & gemcitabine in treatment arm 2

INTERVENTIONS:
Drug: Atu027 & gemcitabine in lead in safety period — Subjects will be treated in a 28-day cycle with Atu027 twice weekly for 4 weeks and gemcitabine once weekly for the first three weeks.
  Arms: Lead in safety period
Drug: Atu027 & gemcitabine in treatment arm 1 — Subjects will be treated in a 28-day cycle with Atu027 and gemcitabine once weekly for three consecutive weeks (on days 1, 8, and 15). During week four no treatment is administered.
  Treatment will be continued in consecutive 28-day cycles until unacceptable toxicity or disease progression occurs.
  Arms: Treatment arm 1
Drug: Atu027 & gemcitabine in treatment arm 2 — Subjects will be treated in a 28-day cycle with gemcitabine once weekly (on days 4, 11, and 18) and Atu027 twice weekly (on days 1, 4, 8, 11, 15, 18, 22, and 25). The 28-day combination cycle is followed by a 28-day gemcitabine monotherapy cycle.
  Treatment will be continued in consecutive 28-day cycles until unacceptable toxicity or disease progression occurs.
  Arms: Treatment arm 2

SUMMARY:
The purpose of the study is to evaluate a new treatment strategy for advanced pancreatic cancer disease by combining the new investigational medicinal product Atu027 with the standard chemotherapeutic gemcitabine. This combination aims at enhancing gemcitabine´s anti-tumor activity with Atu027.

The objectives of this clinical trial are to evaluate safety and activity of two Atu027 schedules in combination with standard gemcitabine treatment in patients with advanced or metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

Lead-in safety period:

* Subjects between the age of 18 and 84 years
* Histologically or cytologically confirmed advanced or refractory cholangiocellular carcinoma, biliary tract cancer, non-small-cell lung carcinoma, duodenal cancer, soft tissue sarcoma, ovarian carcinoma, or another non-pancreatic cancer disease indicated for gemcitabine treatment as determined by the investigator
* Subjects who have previously received chemotherapy and standard curative or palliative care is not available, not effective, or unlikely to be effective
* No option for surgical resection or radiation in curative intent
* Eastern Cooperative Oncology Group (ECOG) performance status assessment of 0 to 2
* Life expectancy of at least 3 months
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Alanine aminotransferase (ALT) ≤3.0 x upper limit of normal (ULN; ≤5 x ULN for subjects with liver metastases)
* Aspartate aminotransferase (AST) ≤3.0 x ULN (≤5 x ULN for subjects with liver involvement with cancer)
* Total bilirubin ≤2.0 x ULN (liver metastasis <5 x ULN)
* Serum creatinine ≤1.5 x ULN
* Adequate bone marrow function: subjects should have an absolute granulocyte count of at least 1,500 (x 10e6/L) and platelet count of 100,000 (x 10e6/L) prior to the initiation of a cycle.
* Prothrombin time-international normalized ratio/partial thromboplastin time (PT-INR/PTT) <1.5 x ULN (subjects who are being therapeutically anti-coagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists). Low-dose aspirin is permitted (≤100 mg daily).
* Women of childbearing potential must have a negative urine pregnancy test at baseline.
* Women of childbearing potential and men must be willing to use highly effective contraceptive methods during the course of the study and 6 months after.
* Subjects must be willing and able (in the opinion of the investigator) to understand the subject information and informed consent form and to comply with the study protocol and procedures.
* Subjects must be willing and able to give written informed consent.

Main part:

* Subjects between the age of 18 and 84 years
* Subjects with locally advanced or metastatic pancreatic adenocarcinoma stage III/IV indicated for gemcitabine treatment as determined by the investigator
* No option for surgical resection or radiation in curative intent
* Histological or cytological documentation of non-hematologic, malignant solid tumor
* At least one measurable lesion or evaluable disease, as per the Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status assessment of 0 to 2
* Life expectancy of at least 3 months
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Alanine aminotransferase (ALT) <=3.0 x upper limit of normal (ULN; <=5 x ULN for subjects with liver metastases)
* Aspartate aminotransferase (AST) <=3.0 x ULN (<=5 x ULN for subjects with liver involvement with cancer)
* Total bilirubin <=2.0 x ULN (liver metastasis <=5 x ULN)
* Serum creatinine <=1.5 x ULN
* Adequate bone marrow function: subjects should have an absolute granulocyte count of at least 1,500 (x 10e6/L) and platelet count of 100,000 (x 10e6/L) prior to the initiation of a cycle.
* Prothrombin time-international normalized ratio/partial thromboplastin time (PT INR/PTT) <1.5 x ULN (subjects who are being therapeutically anti-coagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists). Low-dose aspirin is permitted (≤100 mg daily).
* Women of childbearing potential must have a negative urine pregnancy test at baseline.
* Women of childbearing potential and men must be willing to use highly effective contraceptive methods during the course of the study and 6 months after.
* Subjects must be willing and able (in the opinion of the investigator) to understand the subject information and informed consent form and to comply with the study protocol and procedures.
* Subjects must be willing and able to give written informed consent.

Exclusion Criteria:

Lead-in safety period:

* History of cardiac disease; congestive heart failure >New York Heart Association (NYHA) functional classification system Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; new onset angina within 3 months prior to study entry or unstable angina, or ventricular cardiac arrhythmias requiring anti-arrhythmic therapy
* Poorly controlled diabetes defined as hemoglobin A1c (HbA1c) >=7%
* Poorly controlled hypertension, defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg, despite optimal medical management
* Poorly controlled seizure disorder
* Subjects undergoing renal dialysis
* Known hypersensitivity to the study drugs or active substances or excipients of the preparations
* Pregnant or breast feeding
* Known hepatitis B or C or human immunodeficiency virus (HIV) infection (if documented in the subject's record
* Previous participation in this study
* Current or previous (within 30 days of enrolment) treatment with another investigational drug or participation in another clinical study.
* Subject is a relative of, or staff directly reporting to the investigator.
* Subject is an employee of the sponsor.
* Subject is committed under official or judicial order.
* Any other reason that the investigator considers makes the subject unsuitable to participate

Main part:

* History of cardiac disease; congestive heart failure >New York Heart Association (NYHA) functional classification system Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; new onset angina within 3 months prior to study entry or unstable angina, or ventricular cardiac arrhythmias requiring anti-arrhythmic therapy
* Poorly controlled diabetes defined as hemoglobin A1c (HbA1c) >=8%
* Poorly controlled hypertension, defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg, despite optimal medical management
* Poorly controlled seizure disorder
* Subjects undergoing renal dialysis
* Anticancer chemotherapy or immunotherapy during the study or before first study treatment. Subjects with recurrent disease after adjuvant treatment not progression-free for at least 6 months.
* Radiotherapy to target lesions during study or before study start
* Known hypersensitivity to the study drugs or active substances or excipients of the preparations
* Pregnant or breast feeding
* Known hepatitis B or C or human immunodeficiency virus (HIV) infection (if documented in the subject's record
* Previous participation in this study
* Current or previous (within 30 days of enrolment) treatment with another investigational drug or participation in another clinical study.
* Subject is a relative of, or staff directly reporting to the investigator.
* Subject is an employee of the sponsor.
* Subject is committed under official or judicial order.
* Any other reason that the investigator considers makes the subject unsuitable to participate

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Baseline till follow up visit 1 (18 weeks)
  Time frame will be 18 weeks if patient will be withdrawn after 3 cycles because of disease progression or toxicity.
Subject physical examination | At baseline; later on in 4 week intervals till last follow up visit (1 year);
  Additional time frames in arm 1: 8 days after baseline. Additional time frames in arm 2 and safety cohort (cycle 1 only): 4 and 15 days after baseline.
Measuring of subject vital signs and body weight | At baseline; end of treatment (13 weeks); later on in 4 week intervals till last follow up visit (1 year)
  End of treatment visit will be after 13 weeks only when patient is withdrawn after 3 cycles.
  Additional time frames in arm 1: 8 days after baseline. Additional time frames in arm 2 and safety cohort (cycle 1 only): 4 and 15 days after baseline.
Performance of 12-lead ECG | At baseline; later on in 4 week intervals till end of treatment (13 weeks)
  End of treatment visit will be after 13 weeks only when patient is withdrawn after 3 cycles.
  Additional time frames in arm 1: 8 days after baseline. Additional time frames in arm 2 and safety cohort (cycle 1 only): 4 and 15 days after baseline.
Assessment of clinically significant laboratory parameters outside normal range | At baseline; at end of treatment (week 13 if patient withdrawn after 3 cycles); at follow up visit 1 (week 18 if patient withdrawn after 3 cycles); at each follow up visit till end of trial (1 year)
  Additional time frames in arm 1: During treatment on days 1, 8, 15 of each cycle.
  Additional time frames in arm 2 and safety cohort (cycle 1 only): During treatment on days 1, 4, 8, 11, 15, 18, 22, 25 of each cycle.
Maximum concentration (Cmax), area under the curve (AUC), time to maximum concentration (tmax), and half life (t½) of the Atu027 siRNA single strand (A-strand), and of AtuFect01 and the helper lipid DPyPE | At end of treatment (week 13 if patient withdrawn after 3 cycles); at follow up visit 1 (week 18 if patient withdrawn after 3 cycles)
  Additional time frames in arm 1: During cycles 1 and 2 of treatment on days 1, 8, 15 of each cycle; in cycle 3 and following only on day 1; Additional time frames in arm 2 and safety cohort (cycle 1 only): During the first treatment cycle on days 1, 4, 8, 11, 15, 18; in cycle 3 and following odd numbered cycles only on day 1; in all even numbered cycles no samples are taken.
  Pharmacokinetics will be assessed in subjects of the safety cohort and in the first 4 subjects per treatment arm.

SECONDARY OUTCOMES:
Objective response rate | At baseline and in 8 week intervals till end of trial (1 year)
  Response will be assessed by RECIST Version 1.1 using abdominal magnetic resonance imaging (MRI) or computed tomography (CT) scans.
  An objective response is defined when the overall response is complete response (CR), partial response (PR), or stable disease (SD).
Progression-free survival and overall survival | From baseline in 8 week intervals till end of trial (1 year).
  Progression-free survival and overall survival, based on the objective response definition will be analyzed using Kaplan-Meier methods.
ECOG performance score | At baseline; at end of treatment (13 weeks if patient withdrawn after 3 cycles); at follow up visit 1 (18 weeks if patient withdrawn after 3 cycles); at each following follow up visit till end of trial (1 year)
  Additional time frames: During treatment on day 1 of each cycle.
  The ECOG performance status, and its change from baseline, will be summarized descriptively by visit and treatment arm. The ECOG performance status will also be assessed during the 1 year follow-up period of the study and results including changes to baseline will be summarized.
Biomarker response | At baseline; at day 1 of cycle 3; end of treatment (13 weeks if patient withdrawn after 3 cycles); follow up visit 1 (18 weeks if patient withdrawn after 3 cycles)
  Serum protein markers and circulating microRNA will be analyzed and changes to baseline will be summarized descriptively by treatment arm.
Tumor marker response | At baseline; at end of treatment (13 weeks if patient withdrawn after 3 cycles); at follow up visit 1 (18 weeks if patient withdrawn after 3 cycles); at each following follow up visit till end of trial (1 year)
  Additional time frame: At day 1 of cycle 3 and day 1 of each following second cycle; Tumor markers will be summarized descriptively for each analyzed marker.
Quality of life | At baseline; at day 1 of all cycles except cycle 1; at end of treatment (week 13 if patient withdrawn after 3 cycles)
  Different scales of quality of life assessed with the EORTC questionnaire and their changes from baseline will be summarized descriptively by visit and treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Strumberg, Prof.Dr.med., Principal Investigator — Medizinische Klinik III - Hämatologie/Onkologie Marienhospital Herne
Locations (9):
- Germany (9):
  - Charité - Universitätsmedizin Berlin Charité Centrum für Tumormedizin, Berlin
  - Klinikum Dortmund gGmbH Medizinische Klinik Mitte, Dortmund
  - Universitätsklinikum Freiburg, Innere Medizin II, Freiburg im Breisgau
  - Medizinische Klinik III - Hämatologie/Onkologie Marienhospital Herne, Herne
  - Klinikum Kassel GmbH Medizinischen Klinik IV;Onkologie,, Kassel
  - Klinikum Nürnberg Nord Medizinische Klinik 5, Nuremberg
  - Klinik und Poliklinik für Innere Medizin I Universitätsklinikum Regensburg, Regensburg
  - Klinikum Stuttgart Klinik Hämatologie, Onkologie und Palliativmedizin, Stuttgart
  - Universitätsklinikum Ulm Zentrum für Innere Medizin, Ulm

REFERENCES:
- [Derived] Schultheis B, Strumberg D, Kuhlmann J, Wolf M, Link K, Seufferlein T, Kaufmann J, Feist M, Gebhardt F, Khan M, Stintzing S, Pelzer U. Safety, Efficacy and Pharcacokinetics of Targeted Therapy with The Liposomal RNA Interference Therapeutic Atu027 Combined with Gemcitabine in Patients with Pancreatic Adenocarcinoma. A Randomized Phase Ib/IIa Study. Cancers (Basel). 2020 Oct 26;12(11):3130. doi: 10.3390/cancers12113130. PMID 33114652